CLINICAL TRIAL: NCT01067469
Title: Randomized Phase II Trial of Standard Dose Bevacizumab Versus Low Dose Bevacizumab Plus Lomustine (CCNU) In Adults With Recurrent Glioblastoma Multiforme
Brief Title: Standard Dose Bevacizumab Versus Low Dose Bevacizumab Plus Lomustine (CCNU) for Recurrent Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0597; NCI-2011-00559 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Brain Cancer; Glioblastoma
Keywords: CNS; Central Nervous System; malignant brain tumor; Recurrent Glioblastoma Multiforme; GBM; Bevacizumab; Lomustine; CCNU
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Bevacizumab; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Dose Bevacizumab (Experimental): Bevacizumab 10 mg/kg by vein (IV) over 90 minutes on Days 1, 15, and 29 of 6 week cycle.
  Interventions: Drug: Standard Dose Bevacizumab
- Low Dose Bevacizumab + Lomustine (Experimental): Bevacizumab 5 mg/kg IV over 90 minutes on Day 1 and 22 (every 3 weeks) of 6 week cycle. Lomustine starting dose of 75 mg/m2 administered orally at sleep time on Day 3 of every 6 week cycle.
  Interventions: Drug: Low Dose Bevacizumab; Drug: Lomustine

INTERVENTIONS:
Drug: Standard Dose Bevacizumab — 10 mg/kg by vein (IV) over 90 minutes on Days 1, 15, and 29 of 6 week cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: Standard Dose Bevacizumab
Drug: Low Dose Bevacizumab — 5 mg/kg IV over 90 minutes on Day 1 and 22 (every 3 weeks) of 6 week cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: Low Dose Bevacizumab + Lomustine
Drug: Lomustine — Starting dose of 75 mg/m2 administered orally at sleep time on Day 3 of every 6 week cycle.
  Other Names: CeeNU; CCNU
  Arms: Low Dose Bevacizumab + Lomustine

SUMMARY:
The goal of this clinical research study is to learn if the combination of bevacizumab and lomustine can help to control glioblastoma. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Lomustine is designed to damage the DNA (genetic material of cells) of tumor cells, which may cause the tumor cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being in either group.

* If you are in Group 1, you will receive a higher dose of bevacizumab.
* If you are in Group 2, you will receive lomustine and a lower dose of bevacizumab

Study Drug Administration:

Each treatment cycle is 42 days.

If you are in Group 1:

On Days 1, 15, and 29 of every cycle, you will receive bevacizumab by vein over 90 minutes.

If you are in Group 2:

* On Days 1 and 22 of every cycle, you will receive bevacizumab by vein over 90 minutes.
* On Day 3 of every cycle, you will take lomustine by mouth 1 time a day. You should take lomustine at bedtime 1 hour before or 2 hours after your last meal of the day with 1 cup (about 8 ounces) of water.

Study Visits:

If you are in Group 1 or 2, every 6 weeks:

* You will be asked about any drugs you may be taking and if you have had any side effects.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a neurological exam.
* Your performance status will be recorded.
* You will have an MRI scan.
* If you are on anti-seizure drugs, blood (about 1 teaspoon) will be drawn to measure the amount of anti-seizure drugs in your blood.

If you are in Group 1:

* During Weeks 1-6, blood (about 3 teaspoons) drawn for routine tests 1 time a week.
* After Week 6, blood (about 3 teaspoons) will be drawn for routine tests every 2 weeks.
* On Weeks 2, 4, and 6, and then every 6 weeks after that, urine will be collected to check your kidney function.

If you are in Group 2:

* During Weeks 1-6, blood (about 3 teaspoons) drawn for routine tests 1 time a week.
* After Week 6, blood (about 3 teaspoons) will be drawn for routine tests every 3 weeks.
* On Weeks 3 and 6, and then every 6 weeks after that, urine will be collected to check your kidney function.

Length of Study:

You may stay on study treatment of lomustine and/or bevacizumab for up to 1 1/2 years. After that, you may continue taking bevacizumab for as long as the study doctor thinks it is in your best interest. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

End of Study Treatment Visit:

After you are off study treatment, you will have an end of study treatment visit. At this visit, you may have some or all of the following tests and procedures performed:

* You will be asked about any drugs you may be taking and if you have had any side effects.
* You will have physical exam, including measurement of your vital signs and weight.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have a neurological exam.
* Your performance status will be recorded.

Long-Term Follow-up:

After the end of study treatment visit, the study staff will call you every 3 months to check how you are doing. Each phone call will take about 5 minutes.

This is an investigational study. Bevacizumab and lomustine are FDA approved drugs and commercially available for the treatment of brain tumors. The use of these drugs in this combination is investigational.

Up to 102 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age >/= 18 years
3. Histologically confirmed glioblastoma in first, second or third relapse. A pathology report constitutes adequate documentation of histology for study inclusion. Subjects with an initial diagnosis of a lower grade glioma are eligible if a subsequent biopsy is determined to be glioblastoma. The amount of prior systemic therapy for this population is, nevertheless, restricted to three regimens, with one including temozolomide.
4. Radiographic demonstration of disease progression following prior therapy
5. Bi-dimensionally measurable disease with a minimum measurement of 1 cm (10 mm) in one diameter on MRI performed within 14 days prior to registration (Day 1). Baseline MRIs for subjects who underwent salvage surgery after first or second relapse must be obtained >/= 4 weeks after the procedure. If receiving corticosteroids, subjects must be on a stable or decreasing dose of corticosteroids for >/= 5 days prior to baseline MRI.
6. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply: 1) They have recovered from the effects of surgery. 2) Evaluable or measurable disease following resection of recurrent tumor is not mandated for eligibility into the study. 3) To best assess the extent of residual measurable disease post-operatively, a MRI should be done no later than 96 hours in the immediate post-operative period or 4-6 weeks post-operatively. .
7. An interval of >/= 4 weeks since surgical resection is required prior to starting protocol therapy.
8. Prior standard radiation for glioblastoma
9. Prior chemotherapy: All first-relapse subjects must have received temozolomide. All second- and third-relapse subjects must have received temozolomide. Patients may not have received prior nitrosoureas.
10. Recovery from the effects of prior therapy, including the following: Four weeks from cytotoxic agents (3 weeks from procarbazine, 2 weeks from vincristine); Four weeks from any investigational agent; One week from non-cytotoxic agents(eg accutane, thalidomide); Eight weeks from radiotherapy to minimize the potential for MRI changes related to radiation necrosis that might be misdiagnosed as progression of disease, or 4 weeks if a new lesion, relative to the pre-radiation MRI, develops that is outside the primary radiation field; Patients may have had gliadel wafers during their original surgery but they must be >/= 9 months post their original surgery date.
11. Prior therapy with gamma knife or other focal high-dose radiation is allowed, but the subject must have subsequent histologic documentation of recurrence or positron emission tomography (PET) or MR Spectroscopic documentation of tumor, unless the recurrence is a new lesion outside the irradiated field
12. Patients must have adequate bone marrow function (WBC >/= 3,000/µl, absolute neutrophil count (ANC) >/= 1,500/mm^3, platelet count of >/= 100,000/mm^3, and hemoglobin >/= 10 gm/dl), adequate liver function (SGPT < 3 times normal and alkaline phosphatase < 2 times normal, bilirubin <1.5 mg/dl), adequate renal function (creatinine </= 1.5 mg/dL or creatinine clearance >/= 60 cc/min/1.73 m^2) and a urine protein:creatinine ratio of </=1 before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
13. Patients must have a Karnofsky performance status (KPS) equal or greater than 60
14. Use of an effective means of contraception in males and in females of childbearing potential. Women of childbearing potential must have a negative β-human chorionic gonadotropin (HCG) pregnancy test documented within 14 days prior to registration. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
15. Ability to comply with study and follow-up procedures
16. Patients receiving treatment with other antiepileptic medications will not be excluded. Patients should preferably be treated with non-enzyme inducing anti-epileptic medications to avoid any potential interactions with lomustine. However, the use of non-enzyme inducing anti-epileptic medications is not mandatory. If enzyme-inducing antiepileptic drugs are used, monitoring of drug levels should be considered, as considered clinically appropriate by the treating physician.
17. Patients on the following medications will be included: Anticoagulants/Anti-platelets: Patients on stable dose anticoagulants (e.g. warfarin, low molecular-weight heparin) and in-range international normalized ratio (INR) (2-3) are eligible. Patients are allowed to take aspirin, clopidogrel, ticlopidine, Aggrenox, ibuprofen and other NSAIDS.
18. Patients must be willing to forego other cytotoxic and non-cytotoxic drug therapy against the tumor while enrolled in the study.
19. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

Exclusion Criteria:

1. Prior treatment with anti-angiogenesis (eg bevacizumab, sorafenib, sunitinib) agent or nitrosurea (eg. lomustine, carmustine, nimustine).
2. Prior treatment with polifeprosan 20 with carmustine wafer except for the patients with gliadel wafers >/= 9 months post their original surgery date.
3. Patients must not have received any investigational agents within 28 days prior to commencing study treatment.
4. Prior intracerebral agents
5. Need for urgent palliative intervention for primary disease (e.g., impending herniation)
6. Evidence of recent hemorrhage on baseline MRI of the brain with the following exceptions: (1) Presence of hemosiderin (2) Resolving hemorrhagic changes related to surgery (3) Presence of punctate hemorrhage in the tumor
7. Blood pressure of > 140 mmHg systolic and > 90 mmHg diastolic
8. History of hypertensive encephalopathy
9. New York Heart Association (NYHA) Grade II or greater chronic heart failure(CHF)
10. History of myocardial infarction or unstable angina within 6 months prior to Day 1
11. History of stroke or transient ischemic attack within 6 months prior to study enrollment
12. Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 1
13. Evidence of bleeding diathesis or coagulopathy or INR >1.5 unless on a stable dose of anticoagulation therapy. History of significant bleeding disorder unrelated to cancer, including: (1) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease) (2) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies) (3) Ongoing or recent (</= 3 months) significant gastrointestinal bleeding
14. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
15. History of intracerebral abscess within 6 months prior to Day 1
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study
17. Minor surgical procedures (excluding placement of a vascular access device), stereotactic biopsy, fine needle aspirations, or core biopsies within 7 days prior to Day 1
18. Serious non-healing wound, ulcer, or bone fracture
19. Pregnancy (positive pregnancy test) or lactation
20. Known hypersensitivity to any component of bevacizumab
21. History of any other malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
22. Pregnant or nursing females
23. Unstable systemic disease, including active infection, uncontrolled hypertension, or serious cardiac arrhythmia requiring medication
24. Subjects unable to undergo an MRI with contrast
25. Patients with a known allergy to bevacizumab, or a known allergy to nitrosoureas (eg. lomustine, carmustine, nimustine) will be excluded
26. Patient must be able to tolerate the procedures required in this study including periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study. Inability to comply with protocol or study procedures (for example, an inability to swallow tablets) will be an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John DeGroot, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2010 to January 2015. All recruitment done The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 83 participants enrolled 12 were screen failures and therefore never assigned to treatment arms.
Groups:
- Low Dose Bevacizumab + Lomustine: Bevacizumab 5 mg/kg IV over 90 minutes on Day 1 and 22 (every 3 weeks) of 6 week cycle. Lomustine starting dose of 90 mg/m2 administered orally at sleep time on Day 3 of every 6 week cycle. Due to hematologic toxicities, the starting dose was reduced to 75 mg/m2.
Period: Overall Study
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
Started | 36 | 35
90 mg/m^2 | 0 | 12
75 mg/m^2 | 0 | 21
Completed | 36 | 33
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Median (Full Range); unit: years] — Age at diagnosis
  years | 56 [29 to 75] | 56 [24 to 72] | 56 [24 to 75]
Age, Customized [Count of Participants; unit: Participants]
  <=50 years | 13 | 13 | 26
  >50 years | 23 | 22 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 36 | 35 | 71
Region of Enrollment [Number; unit: participants]
  United States | 36 | 35 | 71
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — KPS index scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities.
  Participants
    60-80 | 13 | 11 | 24
    90-100 | 23 | 24 | 47
# Previous recurrence [Count of Participants; unit: Participants] — Recurrence of cancer prior to treatment on study.
  Participants
    1st | 24 | 25 | 49
    2nd | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Participants with no disease progression as measured by magnetic resonance imaging (MRI) scans. Participants followed by MRI scans, as used for baseline tumor measurements, and removed from study if progression is documented after any cycle of treatment. PFS determined from date of registration in the trial and not date of randomization into chemotherapy arms (i.e. after surgery for resection of recurrent tumor).
Time Frame: Documented from the date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
Number analyzed (Participants) | 36 | 33
months | 4.11 [2.96 to 5.55] | 4.34 [2.96 to 8.34]

2. Secondary Outcome: Radiographic Response (RR)
Description: Definition of Modified Radiographic Response Assessment Criteria for Glioblastoma (GBM) . Complete, Partial, Progressive Disease and Stable Disease. Radiographic response determined in comparison to the tumor measurements obtained at baseline (post-radiation scan will be baseline for newly diagnosed GBM and pre-treatment scans will be the baseline for recurrent GBM) for determination of response, and the smallest tumor measurement at either pre-treatment baseline or following initiation of therapy for determining progression.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
Number analyzed (Participants) | 36 | 33
Participants
  Complete Response | 0 | 0
  Partial Response | 11 | 3
  Progressive Disease | 11 | 9
  Stable Disease | 13 | 19

3. Secondary Outcome: 6-month Progression-free Survival (PFS-6)
Description: as for outcome 1
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
Number analyzed (Participants) | 36 | 33
percentage of participants | 23.6 [12.9 to 43.3] | 36.4 [23.3 to 57.1]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival(OS) is defined: Time of presentation to date of death or censored at last follow-up date
Time Frame: through study completion, an average of 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
Number analyzed (Participants) | 36 | 33
Months | 8.3 [6.42 to 11.58] | 9.6 [6.26 to 16.73]

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from randomization to time of progressive disease
Time Frame: Up to One year
Population: Data were not collected for the outcome for Time to Progression (TTP)
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Summary of Treatment Related Toxicities
Description: Adverse Events grade 3 and 4 hematologic toxicities reported in safety profile of bevacizumab (Avastin) in combination with Lomustine in patients with recurrent glioblastoma using Common Terminology Criteria for Adverse Events (CTCAE) version 3.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
Number analyzed (Participants) | 36 | 33
Participants | 0 | 24

ADVERSE EVENTS:
Time Frame: Adverse event data collected every six weeks after baseline, up to one year (52 weeks).
Arm/Group | Standard Dose Bevacizumab | Low Dose Bevacizumab + Lomustine
All-Cause Mortality (participants affected / at risk) | 6/36 | 1/33
Serious Adverse Events (participants affected / at risk) | 9/36 | 9/35
Other Adverse Events (participants affected / at risk) | 26/36 | 23/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Bevacizumab (N=36) | Low Dose Bevacizumab + Lomustine (N=35)
CNS Ischemia (Nervous system disorders) | 2 (2) | 0 (0)
CNS Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 2 (2) | 2 (2)
Vessel injury - artery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle weakness - generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Perforation, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mental status change (Nervous system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Thrombus, embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Bevacizumab (N=36) | Low Dose Bevacizumab + Lomustine (N=35)
alk phos (Metabolism and nutrition disorders) | 4 (4) | 7 (18)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 6 (11)
ALT/SGPT (Metabolism and nutrition disorders) | 14 (35) | 11 (43)
anorexia (Gastrointestinal disorders) | 6 (14) | 13 (29)
AST/SGOT (Metabolism and nutrition disorders) | 5 (10) | 10 (31)
ataxia (Nervous system disorders) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes